CLINICAL TRIAL: NCT05159583
Title: Commercializing In-Home Supportive Technology for Dementia Caregivers
Brief Title: In-Home Technology for Caregivers of People With Dementia and Mild Cognitive Impairment: Rural Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: People Power Company (Industry); National Institute on Aging (NIA) (NIH); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Robert Levenson, Professor of the Graduate School, Department of Psychology, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1247267250000-1; 2SB1AG059458-04A1 (NIH)
Record Dates: First submitted 2021-12-02; First posted 2021-12-16 (Actual); Results first posted 2025-01-07 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Dementia; Mild Cognitive Impairment; Alzheimer Disease
Keywords: Caregivers; Dementia; Mild Cognitive Impairment; In-Home Technology; Alzheimer's disease; Technology; Rural
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Participants are randomly assigned to treatment arms by People Power. Identical systems are self-installed by caregivers in all homes regardless of treatment arm. Initiating the features of the system appropriate to the assigned treatment arm is done remotely by a member of the People Power staff following the installation. All participants complete the same questionnaires at the same intervals.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-Home Technology System (Experimental): The full system [(a) 1 advanced gateway with a dual-SIM cellular connection to communicate/control the equipment; (b) 5 indoor motion sensors; (c) 3 door/cabinet entry sensors; (d) 1 water leak sensor; (e) 1 "call for help" button; (f) 2 motion-activated LED night lights; (g) 2 Vayyar fall detection and sleep quality sensors] will be self-installed by 60 rural caregivers in their homes. Monitoring of sensors, provision of warnings, messaging, and social networking features will be activated remotely for those participants who have been randomly assigned to this arm. Participation will extend over a 6 month period with questionnaires (e.g., health and well-being) administered 3 times (at the time of installation and every 3 months thereafter).
  Interventions: Device: In-Home Technology System
- Limited In-Home Technology System (Sham Comparator): The full system [(a) 1 advanced gateway with a dual-SIM cellular connection to communicate/control the equipment; (b) 5 indoor motion sensors; (c) 3 door/cabinet entry sensors; (d) 1 water leak sensor; (e) 1 "call for help" button; (f) 2 motion-activated LED night lights; (g) 2 Vayyar fall detection and sleep quality sensors] will be self-installed by 60 rural caregivers in their homes. Only monitoring of the water leak sensor and associated warnings will be activated remotely for those participants who have been randomly assigned to this arm.
  Interventions: Device: Limited In-Home Technology

INTERVENTIONS:
Device: In-Home Technology System — Intelligent bots monitor the in-home sensors, learn typical patterns, and provide caregivers with text messages and alerts via cell phone when worrisome behaviors occur. Caregivers are able to: (a) select services (e.g., warnings for falls, wandering, late night activity); (b) access daily reports (summaries of daily activities that can also be shared with health care providers); and (c) obtain support (e.g. Caregiver Support Groups that connect caregivers with knowledgeable experts and other caregivers, Caregiver Events that provide virtual meetings about relevant topics, and Trusted Circle task management to distribute the caregiving work load).
  Arms: In-Home Technology System
Device: Limited In-Home Technology — Intelligent bots monitor the in-home water leak sensor and provide caregivers with text messages and alerts via cell phone when worrisome conditions occur.
  Arms: Limited In-Home Technology System

SUMMARY:
This study aims to develop, evaluate, and commercialize an in-home supportive technology that is designed to alleviate anxiety, burden, and loneliness in spousal and familial caregivers of individuals with Alzheimer's disease, other dementias, or mild cognitive impairment in rural homes.

DETAILED DESCRIPTION:
This study aims to develop, refine, evaluate, and commercialize a hardware/software system designed to integrate in-home sensors and devices, Internet-of-Things technologies (i.e., devices that can be controlled and communicated with via the internet), and social networking to create a more safe and supportive home environment for caregivers and people who have Alzheimer's disease, other dementias, or mild cognitive impairment. The system monitors troublesome behaviors in people with dementia or mild cognitive impairment (e.g., wandering), and targets mechanisms (e.g., worry, social isolation) thought to link behavioral symptoms in people with dementia or mild cognitive impairment with adverse caregiver outcomes (declines in health and well-being). The system is designed to minimize demands on caregivers' limited time and energy and to provide a platform for data collection that can be used by researchers and care professionals.

Hypotheses:

1. Rural caregivers in the active treatment condition will have better health and well-being (i.e., less caregiver depression, anxiety, loneliness, and burden) and higher user satisfaction compared to those in the control condition.
2. The magnitude of the difference in health and well-being and user satisfaction for rural caregivers in the active treatment condition compared to those in the control condition will increase over time (reflecting additional bot learning and ability to adjust to changing caregiver needs).
3. In the active treatment condition, greater utilization of features (e.g., selecting and receiving warnings, obtaining daily reports, accessing social support services) will be associated with better caregiver health and well-being and higher user satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers are fluent/literate in English
* Caregivers currently reside in the United States with spouse/family member who has received a medical diagnosis of Alzheimer's disease, other dementia, or mild cognitive impairment
* Caregivers live in rural areas (using Rural-Urban Commuting Area Codes data)
* Caregivers primarily use a smartphone (e.g., iPhone, Android)

Exclusion Criteria:

* Caregivers providing care for individuals with known non-neurodegenerative conditions affecting behavior and cognition
* Caregivers providing care for individuals with longstanding Axis I psychiatric disorder
* Caregivers providing care for individuals with metabolic disorder or major organ dysfunction
* Caregivers providing care for individuals with alcohol abuse or dependence (within 5 years of dementia onset)
* Caregivers providing care for individuals with head trauma with loss of consciousness greater than 30 minutes
* Caregivers providing care for individuals with contraindications to MRI imaging
* Caregivers providing care for individuals with large confluent white matter lesions
* Caregivers providing care for individuals with significant systemic medical illness
* Caregivers providing care for individuals who use a medication likely to affect central nervous system functions adversely

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Levenson, Ph.D., Study Director — University of California, Berkeley
Locations (1):
- University of California, Berkeley, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Because health and other protected data are involved, we need to consult with our institutional review board and other collaborators concerning which data can be shared.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Chen KH, Wells JL, Otero MC, Lwi SJ, Haase CM, Levenson RW. Greater Experience of Negative Non-Target Emotions by Patients with Neurodegenerative Diseases Is Related to Lower Emotional Well-Being in Caregivers. Dement Geriatr Cogn Disord. 2017;44(5-6):245-255. doi: 10.1159/000481132. Epub 2017 Dec 8. PMID 29216633
- [Background] Lwi SJ, Ford BQ, Casey JJ, Miller BL, Levenson RW. Poor caregiver mental health predicts mortality of patients with neurodegenerative disease. Proc Natl Acad Sci U S A. 2017 Jul 11;114(28):7319-7324. doi: 10.1073/pnas.1701597114. Epub 2017 Jun 27. PMID 28655841
- [Background] Otero MC, Levenson RW. Lower Visual Avoidance in Dementia Patients Is Associated with Greater Psychological Distress in Caregivers. Dement Geriatr Cogn Disord. 2017;43(5-6):247-258. doi: 10.1159/000468146. Epub 2017 Apr 11. PMID 28395276
- [Background] Brown CL, Lwi SJ, Goodkind MS, Rankin KP, Merrilees J, Miller BL, Levenson RW. Empathic Accuracy Deficits in Patients with Neurodegenerative Disease: Association with Caregiver Depression. Am J Geriatr Psychiatry. 2018 Apr;26(4):484-493. doi: 10.1016/j.jagp.2017.10.012. Epub 2017 Dec 27. PMID 29289452

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Note that outcomes are only assessed regarding caregiver health and well-being. Patients did not provide any information; therefore, all information reported for demographics and measures is only regarding caregivers.
Groups:
- In-Home Technology System: The full system [(a) 1 advanced gateway with a dual-SIM cellular connection to communicate/control the equipment; (b) 5 indoor motion sensors; (c) 3 door/cabinet entry sensors; (d) 1 water leak sensor; (e) 1 "call for help" button; (f) 2 motion-activated LED night lights; (g) 2 Vayyar fall detection and sleep quality sensors] will be self-installed by rural caregivers (N=60) in their homes. Monitoring of sensors, provision of warnings, messaging, and social networking features will be activated remotely for those participants who have been randomly assigned to this arm. Participation will extend over a 6 month period with questionnaires (e.g., health and well-being) administered 3 times (at the time of installation and every 3 months thereafter).
  In-Home Technology System: Intelligent bots monitor the in-home sensors, learn typical patterns, and provide caregivers with text messages and alerts via cell phone when worrisome behaviors occur. Caregivers are able to: (a) select services (e.g., warnings for falls, wandering, late night activity); (b) access daily reports (summaries of daily activities that can also be shared with health care providers); and (c) obtain support (e.g. Caregiver Support Groups that connect caregivers with knowledgeable experts and other caregivers, Caregiver Events that provide virtual meetings about relevant topics, and Trusted Circle task management to distribute the caregiving work load).
- Limited In-Home Technology System: The full system [(a) 1 advanced gateway with a dual-SIM cellular connection to communicate/control the equipment; (b) 5 indoor motion sensors; (c) 3 door/cabinet entry sensors; (d) 1 water leak sensor; (e) 1 "call for help" button; (f) 2 motion-activated LED night lights; (g) 2 Vayyar fall detection and sleep quality sensors] will be self-installed by rural caregivers (N=60) in their homes. Only monitoring of the water leak sensor and associated warnings will be activated remotely for those participants who have been randomly assigned to this arm.
  Limited In-Home Technology: Intelligent bots monitor the in-home water leak sensor and provide caregivers with text messages and alerts via cell phone when worrisome conditions occur.
Period: Overall Study
Arm/Group | In-Home Technology System | Limited In-Home Technology System
Started | 8 | 7
Completed | 6 | 4
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | In-Home Technology System | Limited In-Home Technology System | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (6.14) | 72.14 (11.96) | 71.6 (8.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White (non-Hispanic/Latino) | 8 | 7 | 15
Beck Anxiety Inventory [Mean (Standard Deviation); unit: units on a scale] | 5.5 (6.59) | 10.57 (7.14) | 7.87 (7.11)
Zarit Burden Inventory [Mean (Standard Deviation); unit: units on a scale] | 20.13 (14.08) | 20.71 (8.32) | 20.4 (11.36)
Satisfaction with Life [Mean (Standard Deviation); unit: units on a scale] | 19.5 (10.58) | 20.71 (6.95) | 20.07 (8.78)
Center for Epidemiologic Studies Depression Scale [Mean (Standard Deviation); unit: units on a scale] | 16.13 (13.89) | 17.71 (10.84) | 16.87 (12.14)

OUTCOME MEASURES:

1. Primary Outcome: 3 Months Assessment for Center for Epidemiological Studies Depression Scale (CES-D)
Description: Questionnaire to measure depression (Radloff, 1977). 20 items are rated on a 0-3 scale and summed (range = 0-60). There are no subscales. Higher scores represent worse outcomes. The clinical cut-off is usually set at a score of 16.
Time Frame: 3 months after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- In-Home Technology System: The full system [(a) 1 advanced gateway with a dual-SIM cellular connection to communicate/control the equipment; (b) 5 indoor motion sensors; (c) 3 door/cabinet entry sensors; (d) 1 water leak sensor; (e) 1 "call for help" button; (f) 2 motion-activated LED night lights; (g) 2 Vayyar fall detection and sleep quality sensors] will be self-installed by 60rural caregivers in their homes. Monitoring of sensors, provision of warnings, messaging, and social networking features will be activated remotely for those participants who have been randomly assigned to this arm. Participation will extend over a 6 month period with questionnaires (e.g., health and well-being) administered 3 times (at the time of installation and every 3 months thereafter).
  In-Home Technology System: Intelligent bots monitor the in-home sensors, learn typical patterns, and provide caregivers with text messages and alerts via cell phone when worrisome behaviors occur. Caregivers are able to: (a) select services (e.g., warnings for falls, wandering, late night activity); (b) access daily reports (summaries of daily activities that can also be shared with health care providers); and (c) obtain support (e.g. Caregiver Support Groups that connect caregivers with knowledgeable experts and other caregivers, Caregiver Events that provide virtual meetings about relevant topics, and Trusted Circle task management to distribute the caregiving work load).
Arm/Group | In-Home Technology System | Limited In-Home Technology System
Number analyzed (Participants) | 7 | 5
units on a scale | 17.71 (14.17) | 18.6 (12.7)

2. Primary Outcome: 6 Months Assessment for Center for Epidemiological Studies Depression Scale (CES-D)
Description: as for outcome 1
Time Frame: 6 months after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In-Home Technology System | Limited In-Home Technology System
Number analyzed (Participants) | 6 | 4
units on a scale | 10.33 (6.22) | 19.75 (10.24)

3. Primary Outcome: 3 Months Assessment for Zarit Burden Interview-Short Form
Description: Questionnaire to measure caregiver burden (Zarit, Reever, & Bach-Peterson, 1980). 12 items are rated on 0-4 scale. Range: 0-48. No subscales. Higher scores represent worse outcomes.
Time Frame: 3 months after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In-Home Technology System | Limited In-Home Technology System
Number analyzed (Participants) | 7 | 5
units on a scale | 20.14 (12.29) | 24.2 (11.78)

4. Primary Outcome: 6 Months Assessment for Zarit Burden Interview-Short Form
Description: as for outcome 3
Time Frame: 6 months after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In-Home Technology System | Limited In-Home Technology System
Number analyzed (Participants) | 6 | 4
units on a scale | 19.5 (9.48) | 24 (10.92)

5. Primary Outcome: 3 Months Assessment for Beck Anxiety Inventory (BAI)
Description: Questionnaire to measure anxiety (Beck, Epstein, Brown, & Steer, 1988). 20 items are rated on a 0-3 scale and summed (range= 0-60). Higher scores indicate worse outcomes. There are no subscales. A score greater than 36 is considered to be clinically significant.
Time Frame: 3 months after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In-Home Technology System | Limited In-Home Technology System
Number analyzed (Participants) | 7 | 5
units on a scale | 6.14 (6.04) | 7.8 (5.26)

6. Primary Outcome: 6 Months Assessment for Beck Anxiety Inventory (BAI)
Description: as for outcome 5
Time Frame: 6 months after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In-Home Technology System | Limited In-Home Technology System
Number analyzed (Participants) | 6 | 4
units on a scale | 7.83 (9.13) | 9 (4.4)

7. Primary Outcome: 3 Months Assessment for Satisfaction With Life Scale
Description: Questionnaire measuring overall life satisfaction and well-being (Diener, Emmons, Larsen, & Griffin, 1985). 5 items scored on a 1-7 scale and summed (Range = 5-35). Lower scores indicate worse outcomes. A score of 20 is considered neutral with higher scores considered increasingly more satisfied and lower scores considered increasingly more dissatisfied.
Time Frame: 3 months after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In-Home Technology System | Limited In-Home Technology System
Number analyzed (Participants) | 7 | 5
units on a scale | 20.14 (10.85) | 18.4 (7.23)

8. Primary Outcome: 6 Months Assessment for Satisfaction With Life Scale
Description: as for outcome 7
Time Frame: 6 months after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In-Home Technology System | Limited In-Home Technology System
Number analyzed (Participants) | 6 | 4
units on a scale | 22.33 (9.03) | 15.5 (8.35)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | In-Home Technology System | Limited In-Home Technology System
All-Cause Mortality (participants affected / at risk) | 0/8 | 1/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7

LIMITATIONS AND CAVEATS:
Enrollment was challenging in this rural population. Thirty-eight caregivers initially expressed interest by completing a screening questionnaire but then were unreachable or declined participation before enrolling. Furthermore, 27 caregivers enrolled and completed the first questionnaire packet, but 12 of them discontinued from the study prior to being assigned to one of the two groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT05159583/Prot_002.pdf
  • Statistical Analysis Plan (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT05159583/SAP_003.pdf